CLINICAL TRIAL: NCT01806805
Title: Comparative Study of the Efficiency of Zonisamide in Myoclonus Dystonia: A Monocentric , Randomized in Cross Over and Double Blind Study Versus Placebo Study
Brief Title: Efficacy Trial of Zonisamide for Myoclonus Dystonia
Acronym: EpsilonZêta
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P091104
Record Dates: First submitted 2013-03-06; First posted 2013-03-07 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Myoclonus Dystonia
Keywords: Movement disorder; Myoclonus dystonia; DYT 11; Antiepileptic drugs; Zonisamide; Clinical Trial; Double-mind method
MeSH Terms: conditions — Myoclonic dystonia; Movement Disorders | interventions — Zonisamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zonegran (Experimental): Zonegran / Placebo Zonisamide (Zonegran ®) and its placebo appear under the shape of virgin capsules of size 1. Each drug will be dispensed successively in a box containing blister packs of 14 capsules. For every period (A and B), box will contain 26 blister packs. A phase of progressive increase of doses by stages of 50 mg / week is planned before reaching the fixed dose of 300 in the daytime during 4 weeks. Then, a progressive diminution over two weeks is planned before the stop.
  Interventions: Drug: zonegran; Drug: placebo
- placebo (Placebo Comparator): Placebo /Experimental Zonisamide (Zonegran ®) and its placebo appear under the shape of virgin capsules of size 1. Each drug will be dispensed successively in a box containing blister packs of 14 capsules. For every period (A and B), box will contain 26 blister packs. A phase of progressive increase of doses by stages of 50 mg / week is planned before reaching the fixed dose of 300 in the daytime during 4 weeks. Then, a progressive diminution over two weeks is planned before the stop.
  Interventions: Drug: zonegran; Drug: placebo

INTERVENTIONS:
Drug: zonegran
Drug: placebo

SUMMARY:
Myoclonus Dystonia is a disease in which myoclonus distort the precision of movements and so cause a handicap in the movements of the everyday life. Response to oral medications may be incomplete and surgery may cause operating risk.

Zonisamide is an antiepileptic drug which could bring a therapeutic profit in Myoclonus Dystonia on the severity of the myoclonus.

DETAILED DESCRIPTION:
In "dystonia", the involuntary abnormal movements cause a driving handicap and a change of the quality of life. A particular shape of dystonia, the Myoclonus Dystonia, is characterized by the ascendancy of myoclonias (abrupt and brief movements) associated with the abnormal dystonia. Myoclonus is an additional source of handicap in the movements of the everyday life, because they distort the precision of movements. Response to oral medications may be incomplete and the tolerance poor, such that deep brain stimulation (DBS) surgery is useful for the major forms but it is also an invasive therapeutics which the operating risk is not totally estimated in the absence of controlled study. Therefore, it is necessary to investigate other pharmacological therapeutic tracks which present a good ratio profit / risk.

Zonisamide is usually used in France in the epilepsy's treatment. It showed its efficiency in the progressive myoclonus epilepsy, not only on the seizure but also on the myoclonia. Therefore, it showed its efficiency on post-anoxic and propriospinal myoclonus. So, we make the hypothesis that this medicine could bring a therapeutic profit in the Myoclonus Dystonia.

The aim of this study is to demonstrate the efficiency of the zonisamide on the severity of myoclonus (UMRS) at those patients. The others outcomes are to estimate the impact of the treatment on the myoclonus's neurophysiological characteristics, the dystonia's severity (BFM score), the quality of life (SF-36 and CGI scores), but also to investigate the tolerance of the treatment.

We conducted a randomized, placebo-controlled, double-blind, two-period cross-over design to evaluate the effect on severity of myoclonus in response to placebo or zonisamide (until 300 mg) in 32 patients.

The study includes an evaluation at the beginning and at the end of every period (4 evaluations at all). Each period includes a phase of titration (six weeks) followed by a phase of fixed dose (three weeks). Those two periods are separated by a period of wash-out (3 weeks) preceded by a phase of progressive decrease of doses (two weeks).

ELIGIBILITY:
Inclusion criteria :

* Age >18 and < 60
* Diagnosis of myoclonus dystonia including the isolated myoclonus caused by epsilon-sarcoglycans mutation or deletion.
* Myoclonus present in both hands
* Myoclonus decrease quality of life
* Insufficient efficiency of the benzodiazepine's tolerated maximal dose during one year
* Agreement to use a medically acceptable method of contraception throughout the study for female of childbearing potential
* Normal physical and neurological examination, except myoclonus dystonia
* No hepatic disease
* No renal disease
* Able to comply with study visits and procedures
* Has voluntarily signed consent form
* Taking no medications or stable doses medication for 4 weeks prior to the Baseline visit

Exclusion criteria :

* Patients who are not enrolled at social security
* Individual who have MMS ≤ 24/30 or patients legally protected or inability to provide an informed consent
* Pregnancy, breast feeding women and women who are of childbearing age and not practicing adequate birth control
* Weight < 40 kg
* history of serious psychiatric illness
* history of renal stones
* history of allergy to sulfonamides
* taking medications : topiramate, rifampicin, ketoconazole, cimetidine

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Measure of the evolution of the severity of myoclonus by a specific scale (UMRS) | from day 0 to week 23

SECONDARY OUTCOMES:
Measure of the evolution of the severity of dystonia by a specific scale (BFM) | from day 0 to week 23
measure of the evolution of the severity of myoclonus by electromyographic recording | from day 0 to week 23

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Roze, Principal Investigator — APHP
Locations (1):
- Pitié salpetriere hospital, Paris, France